CLINICAL TRIAL: NCT05991830
Title: Determination of Inflammatory Markers and Level of Cortical Hyperactivity in Older Adults Undergoing Elective Surgery
Brief Title: Inflammatory Markers and Level of Cortical Hyperactivity
Acronym: IMCH
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Sponsor
Other Study IDs: OAIC: 1311/22
Record Dates: First submitted 2023-08-07; First posted 2023-08-15 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Cognition Disorder
MeSH Terms: conditions — Cognition Disorders | interventions — Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Older adults > 60 years
  Interventions: Procedure: General anesthesia

INTERVENTIONS:
Procedure: General anesthesia — Older adults during elective surgery under general anesthesia with propofol, frontal EEG will recorded and a baseline plasma sample will be taken

SUMMARY:
Alzheimer's disease (AD) is a progressive and fatal neurodegenerative disease that is manifested by severe cognitive impairment mainly from late life (>65 years). Clinical studies have shown that both systemic inflammation and cortical and hippocampal hyperactivity are features present in patients during the early stages of the disease. In this project we will seek to relate the levels of the proinflammatory cytokines interleukin-1beta, interleukin-6 and tumor necrosis factor-alpha with the level of cortical hyperactivity evaluated with the electroencephalographic changes induced by the GABAergic anesthetic propofol in older adults undergoing elective surgery.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a progressive and fatal neurodegenerative disease that is manifested by severe cognitive impairment mainly from late life (>65 years). It is now known that markers of damage begin decades before symptoms can be detected, at the stage called preclinical early AD, which progresses inexorably to mild cognitive impairment and ends in severe Alzheimer's dementia. Clinical studies have shown that both systemic inflammation and cortical and hippocampal hyperactivity are features present in patients during the early stages of the disease, however, they have not been directly related in a clinical context. In this project we will seek to relate the levels of the proinflammatory cytokines IL-1beta, IL-6 and TNF-alpha with the level of cortical hyperactivity evaluated with the electroencephalographic changes induced by the GABAergic anesthetic propofol in older adults undergoing elective surgery. The main goal of this project is to determine the levels of inflammatory markers and cortical hyperactivity in older adults. Methodology: the project is an exploratory observational study of a prospective cohort of patients > 60 years of age who will undergo elective surgery under general anesthesia. In the preoperative period, peripheral venous blood samples will be obtained and stored at -80 ° C and then analyzed by the SIMOA® analyzer, fully automated and digital equipment for performing immunoassays, based on SIMOA® technology, which provide an ultrasensitive signal and / or measurement up to 1000 times greater than conventional immunoassays (in the femtomolar range) of proteins. On the other hand, EEG signal at 128 Hz and other variables from BIS® monitor will be recorded to determine the level of cortical hyperactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Adults over 60 years of age undergoing elective surgery
2. Able to understand and sign an informed consent form

Exclusion Criteria:

1. Diagnosis of other neurological pathologies
2. No active acute or chronic decompensated diseases
3. No severe psychiatric illnesses
4. Propofol allergy

Ages: 60 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Cohort of patients > 60 years of age who will undergo elective surgery under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
MoCA score | Baseline (Day 0)
  Score (0 to 30)

SECONDARY OUTCOMES:
Intraoperative EEG | Intraoperative (Day 0)
  EEG parameters
Aβ40 | Baseline (Day 0)
  Aβ40 plasma concentration
Aβ42 | Baseline (Day 0)
  Aβ42 plasma concentration
GFAP™ | Baseline (Day 0)
  Glial Fibrillary Acidic Protein (GFAP™) plasma concentration
Nf-L | Baseline (Day 0)
  Neurofilament light (Nf-L) plasma concentration

CONTACTS AND LOCATIONS:
Overall Officials: Pedro Lobos, PhD, Principal Investigator — University of Chile; Antonello Penna, MD, PhD, Study Chair — University of Chile
Locations (2):
- Chile (2):
  - Centro de Investigación Cínica Avanzada (CICA), Hospital Clinico de la Universidad de Chile, Santiago, RM
  - Hospital Clinico de la Universidad de Chile, Santiago, RM

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared based on individual requests made directly to study investigators